CLINICAL TRIAL: NCT07337096
Title: Electro-acupuncture Plus PD-1 Inhibitors and Chemotherapy as First-Line Treatment for Metastatic Non-Small Cell Lung Cancer: A Randomized Trial
Brief Title: Electro-Acupuncture in Lung cancER : EALER Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou University of Traditional Chinese Medicine (Other)
Collaborators: The First Affiliated Hospital, Guangzhou University of Traditional Chinese Medicine (Other); Jiangsu Province Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BF2025-340
Record Dates: First submitted 2025-12-09; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Non Small Cell Lung Cancer; Accupuncture; PD-1 Inhibitors
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Acupuncture Therapy; Immunotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture (Experimental): Participants will receive 4 times of electro-acupuncture per cycle during the 4-6 cycle of induction chemotherapy combined with PD-1 inhibitors (16-24 sessions of electro-acupuncture in total).
  Interventions: Other: Acupuncture; Drug: Combination of chemotherapy and immunotherapy
- Sham acupuncture (Placebo Comparator): Participants will receive 4 times of sham acupuncture per cycle during the 4-6 cycle of induction chemotherapy combined with PD-1 inhibitors (16-24 sessions of sham acupuncture in total).
  Interventions: Other: Sham acupuncture; Drug: Combination of chemotherapy and immunotherapy

INTERVENTIONS:
Other: Acupuncture — Acupuncture at Neiguan(PC6), Zhongwan (CV12), Guanyuan (CV 4), Baihui (DU20), Yintang (GV29), combined with electro-acupuncture at Zusanli(ST36), and Sanyinjiao (SP-6).
  Other Names: Electro acupuncture; Acupuncture therapy
  Arms: Acupuncture
Other: Sham acupuncture — Sham acupuncture at Neiguan(PC6), Zhongwan (CV12), Guanyuan (CV 4), Baihui (DU20), Yintang (GV29), combined with sham electro-acupuncture at Zusanli(ST36), and Sanyinjiao (SP-6).
  Other Names: Placebo acupuncture
  Arms: Sham acupuncture
Drug: Combination of chemotherapy and immunotherapy — For patients with non-squamous cell carcinoma: PD-1 inhibitor plus AP regimen chemotherapy (Pemetrexed + Carboplatin or Cisplatin, every 3 weeks) for 4-6 cycles.
  For patients with squamous cell carcinoma: PD-1 inhibitor plus TP or GP regimen chemotherapy (Paclitaxel or Liposomal Paclitaxel + Carboplatin or Cisplatin , nab-paclitaxel + Carboplatin or Cisplatin, Gemcitabine + Carboplatin or Cisplatin, every 3 weeks) for 4-6 cycles.

SUMMARY:
This multicentre, randomized controlled trial evaluates the effect and safety of acupuncture combing with PD-1 inhibitors plus chemotherapy in NSCLC. Participants will be randomly assigned to undergo either acupuncture or sham acupuncture concurrent with the initial four-six cycles of chemotherapy combined with PD-1 inhibitors.

DETAILED DESCRIPTION:
This multicenter, randomized controlled clinical trial designed to evaluate the efficacy and safety of electro-acupuncture (EA) as an adjunctive therapy, combined with PD-1 inhibitors and chemotherapy, as a first-line treatment for advanced NSCLC. This trial plans to enroll 424 patients with advanced NSCLC who are negative for actionable driver gene mutations, including but not limited to EGFR and ALK, and a PD-L1 tumor proportion score (TPS) below 50%. Through a central randomization system, participants will be allocated in a 1:1 ratio to either the EA group or the sham-acupuncture control group. The intervention will be administered concurrently with the induction-phase chemotherapy combined with PD-1 inhibitor therapy, for a total of 4 to 6 cycles.

The primary endpoint is progression-free survival (PFS), defined as the time from randomization to the first documented disease progression or death. Secondary efficacy endpoints include overall survival (OS), objective response rate (ORR), disease control rate (DCR), and duration of response (DoR). The symptom burden and health-related quality of life, will be assessed using the Lung Cancer Symptom Scale (LCSS) and the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) with its lung cancer-specific module (QLQ-LC13). Safety and tolerability will be evaluated based on the incidence, severity, and causality of adverse events, graded according to the Common Terminology Criteria for Adverse Events (CTCAE). Immune-related adverse events (irAEs) will be specifically managed per the NCCN Guidelines for Management of Immunotherapy-Related Toxicities. Efficacy analyses will be performed on the full analysis set (FAS) following the intention-to-treat (ITT) principle. Sensitivity analyses will be conducted on the per-protocol set (PPS) to assess the robustness of the primary findings.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed NSCLC, with AJCC lung cancer TNM stage IV.
2. Tumor proportion score for PD-L1 < 50%.
3. Lacks targetable gene mutations (including but not limited to EGFR mutations or ALK fusions).
4. No prior systemic therapy for advanced NSCLC (including chemotherapy, targeted therapy, or immunotherapy). Patients planned to receive first-line (induction) treatment with ICIs plus chemotherapy are eligible. Patients who have received prior neoadjuvant or adjuvant therapy, or definitive chemoradiotherapy, may be enrolled if provided that disease progression occurred more than 6 months after the completion of the last treatment.
5. ECOG performance status score of 0-2.
6. Age ≥ 18 years.
7. At least one measurable lesion per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
8. Adequate organ function (hematology: ANC ≥ 1500/mcL, PLT ≥ 100,000/mcL, Hb ≥ 9.0 g/dL or ≥ 5.6 mmol/L; renal function: estimated creatinine clearance ≥ 50 mL/min; hepatic function: serum total bilirubin ≤ 1.5 × ULN or total bilirubin > 1.5 × ULN with direct bilirubin ≤ ULN, AST and ALT ≤ 2.5 × ULN ≤ 5 × ULN for patients with liver metastases).
9. Voluntary participation in the study, signed informed consent form, good compliance, and cooperation with follow-up.

Exclusion Criteria:

1. Inability to complete baseline assessments.
2. Pregnant or lactating women, and those with psychiatric, intellectual, or language disorders.
3. Patients with autoimmune diseases or hematologic disorders requiring long-term use of hormones or immunosuppressants.
4. Presence of concurrent primary malignant tumors at other sites.
5. Participation in another investigational drug or device clinical trial within 30 days prior to the planned initiation of study treatment.
6. Known seropositivity for human immunodeficiency virus (HIV), other congenital or acquired immunodeficiencies, or history of organ or stem cell transplantation (including autologous bone marrow or peripheral blood stem cell transplantation).
7. Loss of self-care capacity, or any medical, psychological, or ethical condition that, in the investigator's judgment, could interfere with the patient's ability to complete the study.
8. Active skin infection, ulceration, or lesion at acupuncture point sites that would preclude safe administration of treatment.
9. Implanted cardiac pacemaker or other active implantable electronic medical device.
10. Severe needle phobia that would prevent acceptance of needling procedures required by the study protocol.
11. Receipt of any acupuncture or related needle-based therapy within 6 weeks prior to enrollment.
12. Active pneumonitis, or radiation pneumonitis requiring treatment with systemic corticosteroids.
13. Active infection requiring antimicrobial therapy (antibacterial, antifungal, or antiviral agents) according to clinical guidelines at the time of screening. Enrollment may be reconsidered after the infection has been adequately controlled.
14. Active tuberculosis infection, or any severe or uncontrolled systemic illness, including but not limited to clinically significant neurological conditions (e.g., uncontrolled seizures, dementia), unstable or decompensated respiratory, cardiac, hepatic, or renal disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 424 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years.
  Progression-free survival (PFS) is defined as the time from randomization to the first occurrence of either objective disease progression or death from any cause.

SECONDARY OUTCOMES:
Overall survival | From date of randomization until the date of death from any cause, assessed up to 5 years.
  Overall survival is defined as the time from the date of randomization until death due to any cause
Objective response rate | Through study completion, an average of 3 years.
  Objective response rate (ORR) is defined as the proportion of patients achieving a complete response (CR) or partial response (PR) according to iRECIST or RECIST V.1.1 criteria
Disease control rate | Through study completion, an average of 3 years.
  Disease control rate is determined by the percentage of patients who achieve CR, PR, or SD as defined by iRECIST or RECIST V.1.1 criteria. This encompasses all instances of CR, PR, and SD (CR + PR + SD).
Duration of response | Through study completion, an average of 3 years.
  Duration of response (DoR) is defined, for patients with a confirmed objective response (CR or PR), as the time from the date of the first documented response until the date of first documented disease progression or death from any cause.
Quality of life evaluation | At baseline, on Day 8 of each induction chemotherapy cycle (up to 6 cycles, each cycle is 21 days), and on Day 1 of the first maintenance therapy cycle following completion of the induction phase.
  According to the requirements of European Organisation for Research and Treatment of Cancer-quality of life core questionnaire (EORTC QLQ-C30)/Lung cancer 13 items (LC13), the scoring results of each field of the scale were recorded in CRF. The score of this questionnaire ranges between 1 and 4. The higher score indicates the worse quality of life.
Symptom evaluation | At baseline, on Day 8 of each induction chemotherapy cycle (up to 6 cycles, each cycle is 21 days), and on Day 1 of the first maintenance therapy cycle following completion of the induction phase.
  According to the requirements of Lung cancer symptom scale (LCSS), the scoring results of each field of the scale were recorded in CRF. The score of this questionnaire ranges between 0 and 10. The higher score indicates the worse symptom.

CONTACTS AND LOCATIONS:
Overall Officials: Haibo Zhang, Principal Investigator — Guangdong Provincial Hospital of Traditional Chinese Medicine
Locations (3):
- China (3):
  - Guangdong Provincial Hospital of Chinese Medicine, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou University of Chinese Medicine, Guangzhou, Guangdong
  - Jiangsu Provincial Hospital of Chinese Medicine, Nanjing, Jiangsu

IPD SHARING:
Plan to Share IPD: No
Upon study completion and primary results publication, de-identified individual participant data (IPD) that underlie the reported findings may be made available to qualified researchers upon reasonable request. Any data sharing will be contingent on approval of a detailed research proposal and a signed data access agreement, which will include commitments to using the data only for the approved purpose, to securing the data appropriately, and to destroying or returning the data after analysis completion.Researchers interested in accessing the data should contact the corresponding author or the study sponsor.